CLINICAL TRIAL: NCT05454579
Title: The South-East Asian Transgender Health Cohort
Acronym: SEATrans
Status: Recruiting | Type: Observational
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Other Study IDs: IHRI017
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: HIV; STIs; HCV
Keywords: HIV
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- - 150 HIV-positive participants, both who were diagnosed with HIV infection and new cases.: Newly diagnosed HIV-infected participants will be linked to care to start ART. Known HIV-positive participants will be linked to care if they are not in care already. All HIV-positive participants will undergo viral load and CD4 testing at screening/baseline, and be invited back every 6 months for assessment of adherence, viral load testing, STI testing, FBS and lipid profile. A CD4 count will be repeated at Month 12 and Month 24.
- - 150 HIV-negative participants who are already receiving PrEP or who will accept PrEP.: HIV-negative participants will be offered PrEP. Those who accept PrEP will enroll in the PrEP program in each country, undergo creatinine testing at screening/baseline and be invited back at Month 1, Month 3, and every three months thereafter for HIV testing and assessment of adherence. STI testing, FBS, creatinine and lipid profile will be repeated every 6 months.
- - 150 HIV-negative participants who will refuse PrEP.: HIV-negative participants who do not wish to start PrEP will be invited back at every three months for HIV-testing. STI-testing, FBS and lipid profile will be repeated every 6 months.

SUMMARY:
This is a prospective observational cohort study that will enroll 300 HIV-negative transgender people and 150 transgender people living with HIV from 4 community health centers in Thailand, Vietnam, and the Philippines. Each participant will be followed-up until the completion of 24 months.

DETAILED DESCRIPTION:
This prospective observational cohort study will longitudinally track physical (e.g. HIV/STI, sexual risk behavior, gender affirmation, clinical information, cardiovascular health, medical history) and mental health (e.g. stigma and discrimination, gender-based violence, anxiety, depression); identify biomedical, structural, and psychosocial factors impacting physical and mental health among transgender people; describe the structural barriers to healthcare experienced by transgender people as well as develop the guidance on holistic healthcare policies for transgender people.

ELIGIBILITY:
Inclusion Criteria:

* Thai/Vietnamese/Filipino nationality
* Aged ≥ 18 years old
* Self-identify as a transgender woman or transgender man
* Have signed consent form

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * transgender woman or
  * transgender man
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
New cases of HIV infection in transgender people | 24 months
  Longitudinally evaluate medical conditions in physiology by using self-administered questionnaires (e.g. sexual behavioral risk assessment) and laboratory results of anti-HIV over 24 months of follow-up.
Mental health status in transgender people | 24 months
  Longitudinally evaluate the mental health as well as gender violence, stigma, discrimination, substance use, etc. by using self-administered questionnaires (e.g. mental health assessment, psychosocial assessment) including gender affirmation in primary care (e.g., hormones and/or surgical interventions history).
Structural factors and psychosocial factors that impact the physiology and mental health of transgender people | 24 months
  This is related to no.2 and will be collected by using the same questionnaires of self-administered. After collecting and grouping the data, we will know the structure and psychosocial problems that impact the health care system's access of transgender people.

CONTACTS AND LOCATIONS:
Locations (5):
- Victoria by LoveYourself, Pasay, Manila, Philippines
- Thailand (3):
  - Rainbow Sky Association of Thailand (RSAT), Bangkok, Bangkapi
  - Institute of HIV Research and Innovation, Pathum Wan, Bangkok
  - Tangerine Clinic, Institute of HIV Research and Innovation, Pathum Wan, Bangkok
- Glink Clinics, Ho Chi Minh City (HCMC), Vietnam Glink Clinic HCMC1, Ho Chi Minh City, Thuong Kiet Street, Vietnam